CLINICAL TRIAL: NCT05173974
Title: A Randomized, Single-Blind Clinical Study Assessing the Maximum Maxillary Bite Force When Using Two Novel Denture Adhesives Compared to Using No-Adhesive
Brief Title: A Clinical Study to Evaluate the Maximum Maxillary Bite Force (BF) When Using Two Novel Denture Adhesives Compared to Using No-Adhesive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 218042
Record Dates: First submitted 2021-12-17; First posted 2021-12-30 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Denture Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Negative Control (No Intervention): Denture adhesive will not be used.
- Positive Control (Active Comparator): A single application of 1 gram of Super Poligrip Free denture adhesive will be applied topically to oral tissues via the upper denture.
  Interventions: Device: Super Poligrip Free
- Experimental Denture Adhesive 1 (Experimental): A single application of 1 gram of Experimental Denture Adhesive 1 will be applied topically to oral tissues via the upper denture.
  Interventions: Device: Experimental Denture Adhesive 1
- Experimental Denture Adhesive 2 (Experimental): A single application of 1 gram of Experimental Denture Adhesive 2 will be applied topically to oral tissues via the upper denture.
  Interventions: Device: Experimental Denture Adhesive 2

INTERVENTIONS:
Device: Super Poligrip Free — A single application of 1 gram of Super Poligrip Free will be applied topically to oral tissues via the upper denture.
  Arms: Positive Control
Device: Experimental Denture Adhesive 1 — A single application of 1 gram of Experimental Denture Adhesive 1 will be applied topically to oral tissues via the upper denture.
  Arms: Experimental Denture Adhesive 1
Device: Experimental Denture Adhesive 2 — A single application of 1 gram of Experimental Denture Adhesive 2 will be applied topically to oral tissues via the upper denture.
  Arms: Experimental Denture Adhesive 2

SUMMARY:
The purpose of this study is to investigate the hold properties of two experimental denture adhesives using established maximum incisal BF methodology.

DETAILED DESCRIPTION:
This will be a single-centre, controlled, randomized, single-blind (with respect to the examiner performing the incisal BF measurements), 4-treatment, 4- period, cross-over study to evaluate the maximum maxillary BF in a population of full maxillary denture wearers. A currently marketed denture adhesive will be used as a positive control, whilst use of no adhesive will be employed as a negative control.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A participant with a completely edentulous maxillary arch restored with a conventional maxillary full denture with an acrylic base. The maxillary denture prosthesis must fulfil all of the following:

  1. At least moderately well-fitting (Kapur Index, Olshan Modification: retention score Greater than or equal to (>=)2, stability score >=2) at the Screening (V1) visit,
  2. Is well made (according to the well-made assessment).
* A participant with BF measurements which satisfy all the following criteria:

  1. The qualifying BF measurements (without adhesive) at V1 (Screening) must be less than or equal to (=<) 9lbs.
  2. At least 2 of the 4 qualifying BF measurements (without adhesive) at V1 (Screening) must be reproducible (within +-2lbs).
  3. The Baseline BF measurement (without adhesive) at V2-5 must be <=9lbs.
  4. The Baseline BF measurement (without adhesive) at V2-5 and at least 1 of the 3 practice BF measurements must be within +-2lbs of each other.
* A participant who is dentate in the mandibular arch or has a partial or full denture in the mandibular arch that is:

  1. sufficiently stable, in the opinion of the investigator, to enable the bite force determination to be performed.
  2. well made (according to the well-made assessment).

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GlaxoSmithKline Consumer Healthcare (GSK CH) employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to Visit 1 and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or experimental product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is pregnant (self-reported) or intending to become pregnant over the duration of the study.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant unwilling or unable to comply with the Lifestyle Considerations.
* A participant who is currently taking or has taken a bisphosphonate drug (that is (i.e.), Fosamax, Actonel, Boniva).
* A participant who uses any medication or has a condition (e.g. insulin dependent diabetes) that, in the opinion of the investigator, would interfere with the conduct of the study.
* A participant who has any clinically significant or relevant oral abnormality (for example (e.g.) temporomandibular joint [TMJ] problems or tooth abnormalities) that, in the opinion of the investigator, could affect the BF measurements or participant safety.
* A participant who has any condition or medication which, in the opinion of the investigator, is currently causing xerostomia or which could interfere with the conduct of the study.
* A participant with a recent history (within the last year) of alcohol or other substance abuse.
* A participant with Oral soft tissue (OST) examination findings (at V1) such as stomatitis, open sores, lesions, cavitied caries lesions, redness or swelling which in the opinion of the investigator, could interfere with the conduct of the study.
* A participant who has previously been enrolled in this study.
* A participant who is unable to comply with study requirements and/or who is not able to reliably perform a valid bite at the examiner's discretion.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Health Research Institute Indiana University School of Dentistry, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center in United States of America (USA).
Pre-assignment Details: A total of 52 participants were screened, of which 45 were enrolled (7 screened participants failed to meet the required criteria for study participation). Forty-three participants were randomized to study treatment (2 enrolled participants were not randomized due to lost to follow-up prior to treatment assignment) and 41 participants completed the study.
Groups:
- Experimental Denture Adhesive 1/Negative Control/Positive Control/Experimental Denture Adhesive 2: Participants in this arm received a single oral topical application of 1.00 +- 0.05 gram of Experimental Denture Adhesive 1, followed by Negative Control (No Denture Adhesive), Positive Control (Super Poligrip Free Denture Adhesive) and Experimental Denture Adhesive 2 in Period 1 (visit 2), Period 2 (Visit 3), Period 3 (Visit 4) and Period 4 (Visit 5) respectively. Each treatment period was separated by a wash out period of at least 1 to 28 days. Study products were applied by site study staff, to clean upper denture fit surface in a pattern consistent with product label and application instructions.
- Experimental Denture Adhesive 2/Positive Control/Negative Control/Experimental Denture Adhesive 1: Participants in this arm received a single oral topical application of 1.00 +- 0.05 gram of Experimental Denture Adhesive 2, followed by Positive Control (Super Poligrip Free Denture Adhesive), Negative Control (No Denture Adhesive) and Experimental Denture Adhesive 1 in Period 1 (visit 2), Period 2 (Visit 3), Period 3 (Visit 4) and Period 4 (Visit 5) respectively. Each treatment period was separated by a wash out period of at least 1 to 28 days. Study products were applied by site study staff, to clean upper denture fit surface in a pattern consistent with product label and application instructions.
- Negative Control/Experimental Denture Adhesive 2/Experimental Denture Adhesive 1/Positive Control: Participants in this arm received a single oral topical application of 1.00 +- 0.05 gram of Negative Control (No Denture Adhesive), followed by Experimental Denture Adhesive 2, Experimental Denture Adhesive 1, Positive Control (Super Poligrip Free Denture Adhesive) in Period 1 (visit 2), Period 2 (Visit 3), Period 3 (Visit 4) and Period 4 (Visit 5) respectively. Each treatment period was separated by a wash out period of at least 1 to 28 days. Study products were applied by site study staff, to clean upper denture fit surface in a pattern consistent with product label and application instructions.
- Positive Control/Experimental Denture Adhesive 1/Experimental Denture Adhesive 2/Negative Control: Participants in this arm received a single oral topical application of 1.00 +- 0.05 gram of Positive Control (Super Poligrip Free Denture Adhesive), followed by Experimental Denture Adhesive 1, Experimental Denture Adhesive 2, Negative Control (No Denture Adhesive) in Period 1 (visit 2), Period 2 (Visit 3), Period 3 (Visit 4) and Period 4 (Visit 5) respectively. Each treatment period was separated by a wash out period of at least 1 to 28 days. Study products were applied by site study staff, to clean upper denture fit surface in a pattern consistent with product label and application instructions.
Period: Period 1 (Visit 2, 1 Day)
Arm/Group | Experimental Denture Adhesive 1/Negative Control/Positive Control/Experimental Denture Adhesive 2 | Experimental Denture Adhesive 2/Positive Control/Negative Control/Experimental Denture Adhesive 1 | Negative Control/Experimental Denture Adhesive 2/Experimental Denture Adhesive 1/Positive Control | Positive Control/Experimental Denture Adhesive 1/Experimental Denture Adhesive 2/Negative Control
Started | 11 | 10 | 11 | 11
Completed | 11 | 10 | 11 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (at Least 1 to 28 Days)
Arm/Group | Experimental Denture Adhesive 1/Negative Control/Positive Control/Experimental Denture Adhesive 2 | Experimental Denture Adhesive 2/Positive Control/Negative Control/Experimental Denture Adhesive 1 | Negative Control/Experimental Denture Adhesive 2/Experimental Denture Adhesive 1/Positive Control | Positive Control/Experimental Denture Adhesive 1/Experimental Denture Adhesive 2/Negative Control
Started | 11 | 10 | 11 | 11
Completed | 11 | 10 | 11 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (Visit 3, 1 Day)
Arm/Group | Experimental Denture Adhesive 1/Negative Control/Positive Control/Experimental Denture Adhesive 2 | Experimental Denture Adhesive 2/Positive Control/Negative Control/Experimental Denture Adhesive 1 | Negative Control/Experimental Denture Adhesive 2/Experimental Denture Adhesive 1/Positive Control | Positive Control/Experimental Denture Adhesive 1/Experimental Denture Adhesive 2/Negative Control
Started | 11 | 9 (One participant did not report for Period 2 and directly entered in Period 3 (skipped Period 2).) | 11 | 11
Completed | 11 | 9 | 11 | 10
Not Completed | 0 | 0 | 0 | 1
Not completed — Baseline bite was not eligible | 0 | 0 | 0 | 1
Period: Washout Period 2 (at Least 1 to 28 Days)
Arm/Group | Experimental Denture Adhesive 1/Negative Control/Positive Control/Experimental Denture Adhesive 2 | Experimental Denture Adhesive 2/Positive Control/Negative Control/Experimental Denture Adhesive 1 | Negative Control/Experimental Denture Adhesive 2/Experimental Denture Adhesive 1/Positive Control | Positive Control/Experimental Denture Adhesive 1/Experimental Denture Adhesive 2/Negative Control
Started | 11 | 9 | 11 | 10
Completed | 11 | 9 | 11 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Period 3 (Visit 4, 1 Day)
Arm/Group | Experimental Denture Adhesive 1/Negative Control/Positive Control/Experimental Denture Adhesive 2 | Experimental Denture Adhesive 2/Positive Control/Negative Control/Experimental Denture Adhesive 1 | Negative Control/Experimental Denture Adhesive 2/Experimental Denture Adhesive 1/Positive Control | Positive Control/Experimental Denture Adhesive 1/Experimental Denture Adhesive 2/Negative Control
Started | 11 | 10 (One participant did not report for Period 2 and directly entered in Period 3.) | 11 | 10
Completed | 11 | 10 | 11 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3 (at Least 1 to 28 Days)
Arm/Group | Experimental Denture Adhesive 1/Negative Control/Positive Control/Experimental Denture Adhesive 2 | Experimental Denture Adhesive 2/Positive Control/Negative Control/Experimental Denture Adhesive 1 | Negative Control/Experimental Denture Adhesive 2/Experimental Denture Adhesive 1/Positive Control | Positive Control/Experimental Denture Adhesive 1/Experimental Denture Adhesive 2/Negative Control
Started | 11 | 10 | 11 | 10
Completed | 11 | 10 | 11 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Period 4 (Visit 5, 1 Day)
Arm/Group | Experimental Denture Adhesive 1/Negative Control/Positive Control/Experimental Denture Adhesive 2 | Experimental Denture Adhesive 2/Positive Control/Negative Control/Experimental Denture Adhesive 1 | Negative Control/Experimental Denture Adhesive 2/Experimental Denture Adhesive 1/Positive Control | Positive Control/Experimental Denture Adhesive 1/Experimental Denture Adhesive 2/Negative Control
Started | 11 | 10 | 11 | 10
Completed | 11 | 9 | 11 | 10
Not Completed | 0 | 1 | 0 | 0
Not completed — Baseline bite was not eligible | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-To-Treat (mITT) population: All randomized participants with at least one post baseline assessment of efficacy.
Groups:
- Overall Study Participants: Participants received a single oral topical application of 1.00 +- 0.05 gram of Experimental Denture Adhesive 1, Experimental Denture Adhesive 2, Positive control (Super Poligrip Free Denture Adhesive) to the upper denture or Negative control (No Denture Adhesive) as per randomization schedule. Study products were applied by site study staff, to clean upper denture fit surface in a pattern consistent with product label and application instructions.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 18
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Over Baseline Over 12 Hours (AOB 0-12) to Compare Maximum Incisal Bite Force
Description: Natural logged incisal Bite Force (BF) measurements were performed to analyze the denture dislodgement as measure of denture adhesive hold efficacy. All BF measurements were conducted by an examiner. AOB 0-12 was used to assess the incisal BF and defined as (Area under the Curve [AUC]0-12) divided by 12 minus baseline BF (pounds [lbs]). AUC was calculated from 0 to 12 hours using the trapezoid method; denoted as AUC 0-12. This transformation was carried out to return the measurement to the same scale as the original observation. AOB 0-12 was analyzed for each of the three treatments in comparison to no denture adhesive treatment group. Higher values of AOB 0-12 demonstrate a stronger bite force over time than lower values. Baseline was defined as BF (lbs) recorded at hour 0 (pre-treatment).
Time Frame: Baseline and up to 12 hours
Population: mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- Experimental Denture Adhesive 1: Participants of this arm received a single oral topical application of 1.00 +- 0.05 gram of Experimental Denture Adhesive 1 to the upper denture applied by site study staff, to clean dry denture fit surface in a pattern consistent with product label and application instructions.
- Experimental Denture Adhesive 2: Participants of this arm received a single oral topical application of 1.00 +- 0.05 gram of Experimental Denture Adhesive 2 to the upper denture applied by site study staff, to clean dry denture fit surface in a pattern consistent with product label and application instructions.
- Positive Control: Participants of this arm received a single oral topical application of 1.00 +- 0.05 gram of Positive control (Super Poligrip Free denture adhesive) to the upper denture applied by site study staff, to clean dry denture fit surface in a pattern consistent with product label and application instructions.
- Negative Control: Participants of this arm did not receive any adhesive to apply on upper denture.
Arm/Group | Experimental Denture Adhesive 1 | Experimental Denture Adhesive 2 | Positive Control | Negative Control
Number analyzed (Participants) | 41 | 42 | 42 | 42
lbs | 0.87 (0.80) | 0.69 (0.70) | 0.89 (0.86) | 0.59 (0.71)
Statistical Analysis 1: Comparison: Experimental Denture Adhesive 1 vs Negative Control; Test type: Superiority; p = 0.037, ANCOVA — P-value included Bonferroni adjustment; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.01 to 0.29] — ANCOVA with treatment and period as fixed effects; covariates for participant level baseline (natural logged) and period level baseline (natural logged) minus participant level baseline (natural logged). Participants included as a random effect
Statistical Analysis 2: Comparison: Experimental Denture Adhesive 2 vs Negative Control; Test type: Superiority; p = 0.044, ANCOVA — P-value included Bonferroni adjustment; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.00 to 0.28] — ANCOVA with treatment and period as fixed effects; covariates for participant level baseline (natural logged) and period level baseline (natural logged) minus participant level baseline (natural logged). Participant included as a random effect
Statistical Analysis 3: Comparison: Positive Control vs Negative Control; Test type: Superiority; p = 0.005, ANCOVA — unadjusted P-value was presented; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.06 to 0.30]; ANCOVA with treatment and period as fixed effects; covariates for participant level baseline (natural logged) and period level baseline (natural logged) minus participant level baseline (natural logged). Participants included as a random effect

2. Secondary Outcome: Area Over Baseline at 0.5, 1, 3, 6 And 9 Hours to Compare Maximum Incisal BF
Description: Natural logged incisal BF measurements were performed to analyze the denture dislodgement as measure of denture adhesive hold efficacy. All BF measurements were conducted by an examiner. AOB 0-t was defined as AUC 0-t divided by "t" minus baseline BF (lbs), where "t" is equal to 0.5, 1, 3, 6 and 9 hours. AUC was calculated from 0 to "t" hours using the trapezoid method; denoted as AUC 0-t. This transformation was carried out to return the measurement to the same scale as the original observation. AOB for 0.5, 1, 3, 6 and 9 hours were analyzed using the trapezoid method. AOB 0-0.5, AOB 0-1, AOB 0-3, AOB 0-6, AOB 0-9 were analyzed for each of the three treatments in comparison to no adhesive treatment group. Higher values of AOB demonstrate a stronger bite force over time than lower values. Baseline was defined as BF (lbs) recorded at hour 0 (pre-treatment).
Time Frame: Baseline, at 0.5, 1, 3, 6 and 9 hours
Population: mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Experimental Denture Adhesive 1 | Experimental Denture Adhesive 2 | Positive Control | Negative Control
Number analyzed (Participants) | 41 | 42 | 42 | 42
lbs
  AOB 0-0.5 | 0.40 (0.36) | 0.34 (0.40) | 0.47 (0.48) | 0.26 (0.37)
  AOB 0-1 | 0.64 (0.52) | 0.51 (0.56) | 0.71 (0.65) | 0.40 (0.52)
  AOB 0-3 | 0.84 (0.65) | 0.65 (0.63) | 0.84 (0.74) | 0.54 (0.63)
  AOB 0-6 | 0.86 (0.75) | 0.71 (0.68) | 0.88 (0.82) | 0.58 (0.68)
  AOB 0-9 | 0.85 (0.79) | 0.71 (0.69) | 0.89 (0.85) | 0.58 (0.70)
Statistical Analysis 1: Comparison: Experimental Denture Adhesive 1 vs Negative Control; Test type: Superiority; p = 0.218, ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.04 to 0.17] — Statistical comparison for AOB 0-0.5
Statistical Analysis 2: Comparison: Experimental Denture Adhesive 2 vs Negative Control; Test type: Superiority; p = 0.034, ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [0.01 to 0.21] — Statistical comparison for AOB 0-0.5
Statistical Analysis 3: Comparison: Positive Control vs Negative Control; Test type: Superiority; p = 0.004, ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.05 to 0.25] — Statistical comparison for AOB 0-0.5
Statistical Analysis 4: Comparison: Experimental Denture Adhesive 1 vs Negative Control; Test type: Superiority; p = 0.058, ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.00 to 0.24] — Statistical comparison for AOB 0-1
Statistical Analysis 5: Comparison: Experimental Denture Adhesive 2 vs Negative Control; Test type: Superiority; p = 0.017, ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.03 to 0.27] — Statistical comparison for AOB 0-1
Statistical Analysis 6: Comparison: Positive Control vs Negative Control; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [0.09 to 0.33] — Statistical comparison for AOB 0-1
Statistical Analysis 7: Comparison: Experimental Denture Adhesive 1 vs Negative Control; Test type: Superiority; p = 0.004, ANCOVA; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.06 to 0.30] — Statistical comparison for AOB 0-3
Statistical Analysis 8: Comparison: Experimental Denture Adhesive 2 vs Negative Control; Test type: Superiority; p = 0.010, ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.04 to 0.27] — Statistical comparison for AOB0-3
Statistical Analysis 9: Comparison: Positive Control vs Negative Control; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.07 to 0.31] — Statistical comparison for AOB0-3
Statistical Analysis 10: Comparison: Experimental Denture Adhesive 1 vs Negative Control; Test type: Superiority; p = 0.022, ANCOVA; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [0.02 to 0.29] — Statistical comparison for AOB 0-6
Statistical Analysis 11: Comparison: Experimental Denture Adhesive 2 vs Negative Control; Test type: Superiority; p = 0.011, ANCOVA; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.04 to 0.30] — Statistical comparison for AOB 0-6
Statistical Analysis 12: Comparison: Positive Control vs Negative Control; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.06 to 0.33] — Statistical comparison for AOB 0-6
Statistical Analysis 13: Comparison: Experimental Denture Adhesive 1 vs Negative Control; Test type: Superiority; p = 0.037, ANCOVA; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.01 to 0.27] — Statistical comparison for AOB 0-9
Statistical Analysis 14: Comparison: Experimental Denture Adhesive 2 vs Negative Control; Test type: Superiority; p = 0.013, ANCOVA; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.04 to 0.30] — Statistical comparison for AOB 0-9
Statistical Analysis 15: Comparison: Positive Control vs Negative Control; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.06 to 0.32] — Statistical comparison for AOB 0-9

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious Adverse Events (SAEs), Non-SAEs and Medical Device incidents were collected from immediately after signing of informed consent until 5 days following last administration of the study product (Visit 5 treatment Period 4) (Collected up to 39 days)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A SAE is a particular category of an adverse event where the adverse outcome is serious. Treatment emergent adverse events were presented treatment wise.
Arm/Group | Experimental Denture Adhesive 1 | Experimental Denture Adhesive 2 | Positive Control | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42 | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 6/41 | 3/42 | 4/42 | 3/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Denture Adhesive 1 (N=41) | Experimental Denture Adhesive 2 (N=42) | Positive Control (N=42) | Negative Control (N=42)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oral pruritus (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Gingival injury (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Mouth injury (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT05173974/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT05173974/SAP_001.pdf